CLINICAL TRIAL: NCT06000579
Title: The Effect of Emotional Freedom Technique on Premenstrual Syndrome and Pain in University Students: A Randomized Controlled
Brief Title: The Effect of Emotional Freedom Technique on Premenstrual Syndrome and Pain in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: EMEL EGE (Unknown); KAMİLE ALTUNTUĞ (Unknown); Merve YAZAR (Unknown)
Responsible Party: Principal Investigator, Hafize Dağ Tüzmen, LECTURER, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MrvHfz
Record Dates: First submitted 2023-06-04; First posted 2023-08-21 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Premenstrual Syndrome
Keywords: Emotional Regulation, Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): EFT will be applied to individuals with premenstrual syndrome.
  Interventions: Other: EFT
- Control Group (No Intervention): Individuals in the control group will not be interfered with.

INTERVENTIONS:
Other: EFT — Each student will be asked to voluntarily give their phone number and last menstrual cycle date, and the day will be determined for the first session. Then, the first EFT session will be made by the researchers by calling 14 days before the menstruation date. In the 2nd and 3rd sessions, a total of 3 sessions of EFT will be applied face-to-face by the researchers 14 days before menstruation. After each student completes three menstrual cycles, the researchers will meet with the student and PMSS will be applied as a post-test.
  Arms: Experimental Group

SUMMARY:
PMS is one of the common menstrual disorders affecting many young women, and according to epidemiological data, approximately 75% of women have PMS symptoms and 3-8% have severe PMS symptoms. The prevalence of PMS was different in different countries, with 34% in China , 72% in Turkey , 80% in Pakistan and Jordan. It was detected in the range of 92% in India and 14.3%-74.4% in India. Common premenstrual symptoms include anxiety, lack of concentration, depression, bloating, abdominal cramps, breast tenderness, anger, general body pain, nausea, vomiting, fatigue, decreased concentration, mood swings, headache, anxiety, sleep disturbance, appetite changes. In addition to physical symptoms, studies indicate that individuals reporting PMS experience more stress and anxiety, and their sensitivity to depressive symptoms increases due to hormonal fluctuations. Studies have shown that mindfulness-based cognitive methods are effective in the treatment of mood disorders such as depression. It is thought that modulating many PMS symptoms such as stress and experienced emotional problems through mindfulness-based cognitive methods may be an effective approach for future PMS interventions.

ELIGIBILITY:
Inclusion Criteria:

* Persons with amenorrhea,
* pregnancy,
* menstrual irregularity,
* chronic disease,
* mental disorders,
* psychiatric disorders,
* polycystic ovarian syndrome,
* those who have received training on EFT before and those who have communication problems will not be included in the study.

Exclusion Criteria:

* Female students between the ages of 18-25,
* who scored 111 or higher on the Premenstrual Syndrome Scale (PMSS)
* participated in the study voluntarily will be included in the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premenstrual syndrome is seen in women.
Enrollment: 44 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
premenstrual syndrome and emotional freedom technique | 3 month Wıll Be Followed.
  This outcome is assessed with the premenstrual syndrome scale. The lower the score on the scale, the lower the premenstrual syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YAZAR, Study Chair — merve.yazar@karatay.edu.tr
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No